CLINICAL TRIAL: NCT04933279
Title: Iodine Bioavailability From Different Sources of Dietary Iodine Intake in Human Trail
Brief Title: Bioavailability of Iodine for Natural Kelp and Iodized Salt in Young Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Liu Xiao Bing (Other)
Collaborators: Changzhi Medical College (Other); Shenzhen Center for Chronic Disease Control (Other)
Responsible Party: Sponsor-Investigator, Liu Xiao Bing, Associated Professor, Nationtial Institute of Nutrition and Health, China CDC
Organization: Nationtial Institute of Nutrition and Health, China CDC (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CTR2021000617
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Iodine Bioavailability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium iodide group (Experimental): administrated the subjects with 150 ml - 200 ml iodine-containing spareribs soup delivering ≈ 600 µg or 1200 µg iodine
  Interventions: Dietary Supplement: intrinsic iodine in natural kelp
- Natural kelp group (Experimental): administrated the subjects with a bowl of 45 g or 80 g natural kelp delivering ≈ 600 µg or 1200 µg iodine (intrinsic iodine in natural kelp).
  Interventions: Dietary Supplement: iodine-containg spareribs soup

INTERVENTIONS:
Dietary Supplement: iodine-containg spareribs soup — administrated a 150 ml - 200 ml of iodine-containg spareribs soup delivering ≈ 600 µg or 1200 µg iodine
  Arms: Natural kelp group
Dietary Supplement: intrinsic iodine in natural kelp — administrated 45 g or 80 g natural kelp delivering ≈ 600 µg or 1200 µg iodine (intrinsic iodine). The natural kelp will be approximately produced in an experimental barn feeding supplementary iodine to reach a final iodine intake of ≈ 600 µg or 1200 µg. The iodine intake of natural kelp will be adjusted to the required dose by determing iodine content in the natural kelp.
  Arms: Potassium iodide group

SUMMARY:
Iodine is an essential micronutrient for the production of thyroid hormones and its deficiecny remains a global problem impairing health. The primary source of iodine is the diet via consumption of foods, including cooked foods with iodized salt, dairy products, or naturally abundant seafood. Currently, the recommendation of dietary iodine intake is 150 μg per day in adults who are not pregnant or lactating. The ingestion of iodine or exposure above this threshold is well-tolerated and nearly no health problems are observed. The diets processed and cooked with iodized salt are generally important iodine sources, however, high iodine intake is a result of routine consumption of several kinds of edible algae in coastal regions, with varying contributions depending on the amount of seafood consumed.

Iodine absorption mainly depends on the iodine species in foods and possibly on the iodine status of the individual. Further, there was little available data on iodine absorption or bioavailability from different dietary sources, such as natutal kelp and fortified food with potassium iodide. To our knowledge, inorganic iodide is thought to be absorbed almost completely (over 90%). However, only about two-thirds of some forms of organically-bound iodine are absorbed. The different sources of iodine absorption have not been accurately quantified and compared in humans. Therefore, the purposes of this study were to quantify the iodine absorption of natural kelp in male and female adults and compare with the bioavailability from an iodine water solution (potassium iodide). This stduy will obtain the actual iodine bioavailability and the difference for different source of foods.

This study is a randomized, cross-over design and aims to evaluate the iodine bioavailability (measured using excretion in urine and fece) from different source and administered dose of iodine, such as natural kelp and potassium iodide delivering a dialy iodine intake about 600 µg and 1200 µg. This study will compare and measure to the ingestion of natural kelp and potassium iodide within one subject by three stages: (1) normal iodine intake stage (iodine intake >150 µg/day); (2) intervention stage, a bowl of soup with an extrinsic iodine dose of about 600 µg; or a bowl of natural kelp with a certain iodine content of about 1200 µg potassium iodide.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 25 years; BMI 19-25 kg/m2; Current use of iodized salt at home, adequate iodine nutritional status; Volunteer to participate in and comply with the requirement of study; Signed informed consent.

Exclusion Criteria:

* 1. Having history of thyroid diseases or thyroid dysfunction; 2. Inadequate iodine status (defined as mUIC <100 µg/L or >300 µg/L and assessed during screening by 3-days 24-h urine specimens) 3. Any metabolic, gastrointestinal or chronic disease or chronic use of medications or drug abuse 4. Use of iodine containing supplements within 1 month prior to study start or exposure to iodine-containing X-ray/ computed tomography contrast agent or often use of iodine-containing disinfectants 5. Cannot comply with the requirement of study or cannot delivered the excremental specimens on schedule

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All, half male and half female
Enrollment: 20 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-05-12 (Estimated); Study Completion 2024-05-12 (Estimated)

PRIMARY OUTCOMES:
Urinary Iodine concentration | Time Frame: Day 1th, 2nd, 3rd, 8th, 9th, 10th, 15th, 16th and 17th
  measured by Sandell-Kolthoff method, mikrograms per liter To calculate iodine absorption, excretion and retention.

SECONDARY OUTCOMES:
Sex | 1 day At screening
  male and female
Body Mass Index (BMI) | 1 day At screening
  BMI calculated from measured weight and height.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoguang Yang, Ph.D, Principal Investigator — National Institute of Nutrition and Health, China CDC
Locations (1):
- Changzhi Medical College, Changzhi, Shanxi, China

IPD SHARING:
Plan to Share IPD: No